CLINICAL TRIAL: NCT03511274
Title: Reducing Acquisition of CMV Through Antenatal Education: A Feasibility Study to Assess an Educational Intervention to Prevent Cytomegalovirus Infection in Pregnancy
Brief Title: Reducing Acquisition of CMV Through Antenatal Education
Acronym: RACEFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: University College, London (Other); Kingston University (Other); University of Cambridge (Other); CMV Action (Unknown)
Responsible Party: Principal Investigator, Christine Jones, Honorary Senior Lecturer & Consultant in Paediatric Infectious Diseases, St George's, University of London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PB-PG-0215-36120
Record Dates: First submitted 2017-07-07; First posted 2018-04-27 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Cytomegalovirus Congenital
Keywords: Cytomegalovirus Congenital; CMV; Cytomegalovirus infections
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Intervention Model Description: CMV seronegative pregnant women will be randomised to one of two study arms: treatment as usual or the education intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hygiene based educational film (Experimental): Women randomised to receive the CMV educational intervention will fill in a questionnaire and view the film. The website will also contain interactive information about CMV and how to prevent it. After watching the film and reading the information, women will be asked to fill in a post-intervention questionnaire. The website will be accessible via the participants' own mobile device or computer or dedicated study tablets or computers on-site. Using a web-based intervention, we will be able to monitor use of the educational intervention and also collect data in real time.
  Interventions: Behavioral: Hygiene based educational film
- Treatment as usual (TAU) (No Intervention): Women who are randomised to the TAU group will also be asked to log-on the website. Instead of receiving specific information about prevention of CMV in pregnancy, they will receive information about routine antenatal immunisation. In the UK, the Department of Health recommends that all pregnant women should be offer immunisation against pertussis (whooping cough) and influenza (if pregnant during the influenza session). This will ensure that participants in the TAU arm of the study also derive benefit from the study.

INTERVENTIONS:
Behavioral: Hygiene based educational film — Pregnant women will watch an educational film to increase the awareness of CMV, encourage the adoption of risk reduction behaviours and preventative strategies. The film will include women's views of the risks of CMV infection in pregnancy and how they adopted the preventative strategies.
  Arms: Hygiene based educational film

SUMMARY:
The evidence to date indicates that educational strategies may be effective at reducing antenatal CMV infection, however these have not been tested in the UK.

In phase 1 of the study, the investigators will co-design an educational intervention with pregnant women and families affected by congenital CMV with the aim of reducing the risk of acquisition of CMV in pregnancy. In phase 2 of the study, the investigators will use this educational intervention in a randomised controlled trial (RCT) as part of a feasibility study to generate the data required for the design of a future main RCT. Should the future main RCT show that the educational intervention is effective in reducing the risk of primary CMV infection in pregnancy, the intervention could be rolled out in the National Health Service (NHS). This would have significant benefits to patients and the NHS. No other single cause of congenital defects and long-term developmental disability currently provides greater opportunity for improved outcomes than the prevention of congenital CMV, therefore trials designed to test prevention strategies should be a research priority for the NHS.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) is the most common infection to be contracted before birth (a congenital infection); overall, about 20% of babies infected in this way have permanent health problems, such as hearing loss, learning delay or physical impairments. CMV is not a well-known infection, despite the health problems it can cause. It is actually more common than Down's syndrome or spina bifida. Simple hygiene measures may reduce the risk of catching CMV infection whilst pregnant and therefore also the risk of congenital infection in the infant. In the UK, pregnant women are not routinely counselled about these hygiene measures.

Before a large-scale study can be performed in the UK to determine the effectiveness of an educational intervention in reducing CMV infection in pregnancy, educational materials need to be developed and tested to ensure the feasibility of such a large study.

In this feasibility study, the investigators will work with pregnant women and families affected by CMV to design and produce a short film appropriate for use in the NHS to educate women about these simple hygiene measures (phase 1 of the study). Working in partnership with members of the public will help us ensure the content is relevant, clear and sensitive.The film will subsequently be tested in a study where women are assigned by chance to the educational intervention or to continue with treatment as usual with information about vaccines already recommended within the NHS. This ensures both groups will get some benefit from the study.

This study will enable the investigators to work out the number of pregnant women who are at risk of contracting CMV, how many of these women would agree to take part and to calculate the number of people needed in a future main trial in order to come to a reliable answer. This feasibility study is therefore essential to the design of a large-scale future trial.

ELIGIBILITY:
Inclusion criteria:

• Pregnant women who have children less than 3 years of age booking to St George's Hospital antenatal clinics

Exclusion Criteria:

* Unwilling or unable to give informed consent
* Unwilling or unable to commit to study procedures
* Less than 18 years old

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 878 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Educational intervention development | 3 years
  Develop and refinement of a film-based educational intervention in partnership with pregnant women and families affected by CMV

SECONDARY OUTCOMES:
Proportion of women willing to be screened for CMV | 1 year
  Proportion of women approached who are willing to have antenatal booking blood tested for CMV antibodies to determine serostatus
Proportion of women seronegative at antenatal booking | 1 year
  Proportion of women who have no evidence of previous CMV infection at the time of antenatal booking
Proportion of women with primary CMV infection in the first trimester of pregnancy | 1 year
  Proportion of women who have evidence of primary CMV infection within the first trimester of pregnancy
Proportion of seronegative willing to be randomised to receive educational intervention or treatment as usual | 1 year
  Proportion of seronegative pregnant women willing to participate in feasibility study, which includes randomisation to the educational intervention or treatment as usual
Seroconversion rate | 18 months
  Women will have a second blood sample tested at the end of pregnancy (between 34 weeks and delivery) to determine whether seroconversion has occurred. Seroconversion is the appearance of anti-CMV IgG antibodies in the serum of a person who did not have such antibodies previously. This will be the gold standard evidence for acquisition of primary infection and is the main outcome measure of the future main trial.
Proportion of infants with congenital CMV | 2 years
  The proportion of infants with a positive test for CMV in the first 21 days of life
Measures of adherence | 2 years
  Women in the treatment arm will be asked to a questionnaire to assess their perceptions of adherence to the advice given
Change in knowledge | 2 years
  Women will complete questionnaires before and after the intervention to assess changes in knowledge about CMV
Knowledge of CMV risk reduction measures | 2 years
  Women will complete questionnaires before and after the intervention to assess changes in knowledge about risk reduction measures and self-efficacy towards these
Acceptability of prevention measures | 2 years
  Women will complete questionnaires before and after the intervention to assess the acceptability of prevention measures and to identify barriers to adherence. Interviews will also be carried out to explore these in more depth.
Acceptability of the educational intervention (film) | 2 years
  Perceptions Perceptions and acceptability of the educational intervention will be explored in questionnaires and interviews
Anxiety level | 2 years
  Women in the treatment arm will complete the Perinatal Anxiety Screening Scale and Edinburgh Depression Scale to ensure that study participation does not increase anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Chrissie E Jones, BMBS PhD, Principal Investigator — St George's, University of London
Locations (1):
- St George's, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Calvert A, Vandrevala T, Parsons R, Barber V, Book A, Book G, Carrington D, Greening V, Griffiths P, Hake D, Khalil A, Luck S, Montague A, Star C, Ster IC, Wood S, Heath PT, Jones CE. Changing knowledge, attitudes and behaviours towards cytomegalovirus in pregnancy through film-based antenatal education: a feasibility randomised controlled trial of a digital educational intervention. BMC Pregnancy Childbirth. 2021 Aug 18;21(1):565. doi: 10.1186/s12884-021-03979-z. PMID 34407771